CLINICAL TRIAL: NCT02848352
Title: The Role of Expectations in Experimentally Induced Sadness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016-02v
Record Dates: First submitted 2016-06-29; First posted 2016-07-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Positive placebo group (Experimental): Participants receive a nasal spray that is a placebo. However, they are told that it protects from experiencing negative emotions. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Placebo nasal spray; Other: Film Sequence
- Negative placebo group (Experimental): Participants receive a nasal spray that is a placebo. However, they are told that it sensitizes for experiencing negative emotions. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Placebo nasal spray; Other: Film Sequence
- Placebo control group (Placebo Comparator): Participants receive a nasal spray that is a placebo and are told that it is a placebo. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Placebo nasal spray; Other: Film Sequence
- No-treatment control group (Other): Participants do not receive the nasal spray. Participants watch a film sequence that is supposed to induce sadness.
  Interventions: Other: Film Sequence

INTERVENTIONS:
Other: Placebo nasal spray
  Arms: Negative placebo group; Placebo control group; Positive placebo group
Other: Film Sequence

SUMMARY:
The study aimed at identifying whether different expectations have an impact on experiencing emotions in the form of sadness.

ELIGIBILITY:
Inclusion Criteria:

* fluent in German language

Exclusion Criteria:

* major depression
* current intake of psychotropic medication
* drug intake within the last two weeks
* alcohol consumption within the last twelve hours
* allergic to capsaicin
* allergic to sesame oil
* students in medicine, pharmacy, or psychology in their third year or older

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Sadness (PANAS-X) | Directly after watching the film sequence, no follow-up assessments

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No